CLINICAL TRIAL: NCT06398470
Title: A Feasibility Trial to Evaluate Margin Status During Radical Prostatectomy With En-face Fluorescence Confocal Microscopy (LaserSAFE) Compared to NeuroSAFE
Brief Title: Study to Evaluate a New Method to Detect Residual Tumours During Surgery for Prostate Cancer Using Confocal Microscopy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 159477; 320973 (Other: IRAS number)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Radical prostatectomy; Nerve sparing; Surgical margins; Confocal microscopy
MeSH Terms: conditions — Prostatic Neoplasms; Margins of Excision

STUDY DESIGN:
Intervention Model Description: The investigators aim to recruit a group of 20 patients who will undergo radical prostatectomy as a treatment for prostate cancer. The prostate specimen will be analysed using both techniques, but decisions on how much tissue to resect during surgery will depend on the results of NeuroSAFE.
Masking Description: After LaserSAFE, images are acquired, they will be annotated with the study identifier only. Images will be stored and kept until the end of recruitment. Once all specimens have been evaluated using paraffin analysis, a dedicated meeting with the evaluating pathologist will be carried out. A set of images without any patient identifier will be shown in random order. A purposely built document will allow the pathologist to report the images. This meeting will be repeated with every evaluating pathologist until all images have been analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radical prostatectomy (Other): The patients will undergo radical prostatectomy with nerve sparing decisions based on the results of the NeuroSAFE technique
  Interventions: Diagnostic Test: NeuroSAFE procedure; Diagnostic Test: LaserSAFE procedure

INTERVENTIONS:
Diagnostic Test: NeuroSAFE procedure — Frozen section analysis of the posterolateral surface of the prostate to guide nerve sparing decisions.
Diagnostic Test: LaserSAFE procedure — The LaserSAFE procedure is performed using an FCM called the Histolog® scanner developed by Samantree® which can be placed within the operating room. The Histolog® scanner produces digital images with high, micrometre-range resolution and enables the visualization of tissue microstructures down to the cellular level.
  Other Names: Ex vivo fluorescence confocal microscopy

SUMMARY:
Prostate cancer is the most common solid cancer affecting male patients worldwide. When diagnosed early, it can usually be cured with surgery (radical prostatectomy), but this procedure is associated with side effects such as urinary incontinence and erectile dysfunction. If the nerves that surround the prostate are left intact (nerve-sparing), the risk of developing these side effects decreases. However, since these nerves are in intimate contact with the prostate there is a chance of leaving cancer cells behind, with the subsequent need for additional treatments. Sadly, the current methods surgeons use to select patients who can safely be offered nerve-sparing are not very accurate in predicting where the tumour is extending outside the prostate.

NeuroSAFE is a technique that can inform the surgeon if there are tumour cells on the surface of the prostate and indicate the need for removing more tissue during the same operation. However, it requires a specialised team to process the sample in a reasonable amount of time that does not excessively prolong the surgery. Therefore, many centres are not able to perform it.

A new technology called fluorescence confocal microscopy (LaserSAFE) can be used to examine the surface of the prostate and can identify when cancer is present. Critically, it requires minimal training and resources to produce results in a few minutes and the microscope can be placed in the operating room.

The investigators aim to recruit a group of 20 patients who will undergo radical prostatectomy as a treatment for prostate cancer. The prostate specimen will be analysed using both techniques, but decisions on how much tissue to resect during surgery will depend on the results of NeuroSAFE. This feasibility study will allow us to understand the challenges associated with performing both techniques. This will allow us to plan a larger study to evaluate the accuracy of LaserSAFE.

DETAILED DESCRIPTION:
This trial will be a multi-site, single-blinded, prospective, feasibility study. 20 participants will be recruited from 2 centres that have experience performing the NeuroSAFE technique. Participants will undergo a robotic-assisted radical prostatectomy with nerve-sparing guided by the NeuroSAFE technique. Before the prostate is sent for evaluation the LaserSAFE technique will be used to analyse the corresponding posterolateral surfaces of the prostate. Participating pathologists involved in interpreting the results of NeuroSAFE will be blinded to the LaserSAFE results, to avoid influencing standard patient treatment, management, and progression outcomes after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with operable cT2-T3a N0 M0 prostate cancer.
* Patients who underwent a multiparametric magnetic resonance imaging (MRI) before or after prostate biopsy.
* Medically fit to undergo radical prostatectomy.
* Scheduled for robot-assisted radical prostatectomy with a recommendation against nerve sparing on at least 1 side based on multidisciplinary meetings informed by MRI, biopsy result and clinical factors.
* Ability to read English sufficiently to understand the patient information sheet and to give informed consent.

Exclusion Criteria:

* • Patients who received neo-adjuvant treatment.

  * Patients in whom preoperative imaging shows rectal involvement or seminal vesicle invasion in which nerve sparing is deemed not feasible due to safety concerns.
  * Patients who received previous treatment for prostate cancer: External beam radiotherapy, brachytherapy, focal therapy, chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Feasibility assessment | 8 months
  Evaluate the feasibility of using the LaserSAFE technique to evaluate margin status during radical prostatectomy compared to the NeuroSAFE technique

SECONDARY OUTCOMES:
Concordance | 8 months
  Concordance between LaserSAFE and NeuroSAFE recommendation on secondary resection during radical prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Greg Shaw, Principal Investigator — University College, London
Locations (1):
- University College Hospital at Westmoreland Street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share individual participant data as this is a feasibility study with low number of participants

REFERENCES:
- [Derived] Almeida-Magana R, Mendes LST, Dinneen E, Al-Hammouri T, Haider A, Silvanto A, Freeman A, Roberts N, Dickinson L, So CW, Tandogdu Z, Lamb BW, Mayor N, Winkler M, Ahmed H, Shaw G. The LaserSAFE technique for margin assessment during radical prostatectomy: a feasibility study. BJU Int. 2025 Nov 27. doi: 10.1111/bju.70092. Online ahead of print. PMID 41309506